CLINICAL TRIAL: NCT00995033
Title: A Phase 2B, Multi-Center, Randomized, Double-Blinded, Parallel-Arm , Study to Assess Efficacy and Safety of 3'-Aminomethylnicotine-P. Aeruginosa r-Exoprotein A Conjugate Vaccine (NicVAX®) or Placebo Co-Administered With Varenicline (Champix®) as an Aid in Smoking Cessation
Brief Title: Efficacy and Safety of NicVAX® Co-administered With Varenicline (Champix®)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Nabi Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MEC 08-5-066; ZonMw 40-00812-98-07-004; ZonMw 61200014; Nabi-4508
Record Dates: First submitted 2009-10-06; First posted 2009-10-14 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Smoking Behavior; Smoking Lapse Behavior; Smoking Relapse Behavior
Keywords: Smoking cessation; Smoking lapse behavior; Smoking Relapse behavior; Varenicline; Nicotine conjugate vaccine; Medication effect on smoking lapse behavior
MeSH Terms: conditions — Smoking; Smoking Cessation | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NicVAX conjugate vaccine (Experimental)
  Interventions: Biological: NicVAX vaccine; Drug: Varenicline
- Placebo (Placebo Comparator): Biological
  Interventions: Biological: Placebo; Drug: Varenicline

INTERVENTIONS:
Biological: NicVAX vaccine — NicVAX vaccine given 6 times over 6 months
  Arms: NicVAX conjugate vaccine
Biological: Placebo — Phosphate buffered saline and ALhydrogel of identical appearance to NicVAX; IM in 6 doses over 6 months
  Arms: Placebo
Drug: Varenicline — Days 0-2: 0.5 mg once daily, Days 3-6: 0.5 mg twice daily (morning and evening), Day 7- 84: 1.0 mg twice daily (morning and evening)
  Other Names: Champix; Chantix

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of NicVAX co-administered with varenicline as an aid in smoking cessation over a one-year period in smokers who want to quit smoking.

ELIGIBILITY:
Inclusion Criteria:

* Smokes at least 10 cigarettes per day
* Good general health
* Negative pregnancy test prior to study entry

Exclusion Criteria:

* Prior exposure to NicVAX or any other nicotine vaccine
* Known allergic reaction to alum or any of the components of the vaccine
* Use of systemic steroids, immunosuppressive agents or other medication that might interfere with an immune response
* Cancer or cancer treatment in the last 5 years
* HIV infection
* History of drug or alcohol abuse or dependence within 12 months
* Significant cardiovascular, hepatic, renal, psychiatric and/or respiratory disease
* Previous intolerance to varenicline
* Inability to fulfill all visits for approximately 54 weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 558 (Actual)
Dates: Start 2009-10; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Long term abstinence | one year

SECONDARY OUTCOMES:
Safety, immunogenicity | continuous assessment throughout the one year study duration
Abstinence | continuous assessment throughout the one year study duration
Lapse and relapse rate | continuous assessment throughout the one year study duration
Withdrawal symptoms | continuous assessment throughout the one year study duration

CONTACTS AND LOCATIONS:
Overall Officials: Onno van Schayck, Professor Dr, Principal Investigator — Maastricht University Medical Center
Locations (2):
- Netherlands (2):
  - Maastricht University Medical Center, Maastricht, Limburg
  - Slotervaart Hospital/ Smoking Cessation Clinic, Amsterdam, North Holland

REFERENCES:
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273
- [Derived] Hoogsteder PH, Kotz D, van Spiegel PI, Viechtbauer W, van Schayck OC. Efficacy of the nicotine vaccine 3'-AmNic-rEPA (NicVAX) co-administered with varenicline and counselling for smoking cessation: a randomized placebo-controlled trial. Addiction. 2014 Aug;109(8):1252-9. doi: 10.1111/add.12573. Epub 2014 Jun 3. PMID 24894625
- [Derived] Hoogsteder PH, Kotz D, van Spiegel PI, Viechtbauer W, Brauer R, Kessler PD, Kalnik MW, Fahim RE, van Schayck OC. The efficacy and safety of a nicotine conjugate vaccine (NicVAX(R)) or placebo co-administered with varenicline (Champix(R)) for smoking cessation: study protocol of a phase IIb, double blind, randomized, placebo controlled trial. BMC Public Health. 2012 Dec 6;12:1052. doi: 10.1186/1471-2458-12-1052. PMID 23216646